CLINICAL TRIAL: NCT00676130
Title: Randomized Trial of Trimethoprim-Sulfamethoxazole Versus Placebo Added to Standard Treatment of Uncomplicated Cellulitis in Emergency Department Patients
Brief Title: Study of New Antibiotic Regimen for the Treatment of Uncomplicated Cellulitis in Emergency Department Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Daniel Jay Pallin, MD, MPH, Associate Research Director, Department of Emergency Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007P000414; F8349839
Record Dates: First submitted 2007-12-28; First posted 2008-05-12 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Cellulitis
Keywords: Cellulitis; Bactrim; Trimethoprim Sulfamethoxazole; MRSA; Methicillin-resistant Staphylococcus aureus
MeSH Terms: conditions — Cellulitis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Cephalexin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard therapy (Active Comparator): cephalexin plus placebo
  Interventions: Drug: Cephalexin
- Standard plus anti-CA-MRSA (Experimental): cephalexin plus trimethoprim-sulfamethoxazole
  Interventions: Drug: trimethoprim-sulfamethoxazole; Drug: Cephalexin

INTERVENTIONS:
Drug: trimethoprim-sulfamethoxazole — Weight-based dosing in capsule or suspension form according to the following scale:
  15-19 kg (33-42 lbs): trimethoprim-sulfamethoxazole 40/200 mg four times daily
  20-24 kg (42-53 lbs): trimethoprim-sulfamethoxazole 60/300 mg four times daily
  25-29 kg (53-64 lbs): trimethoprim-sulfamethoxazole 72/360 mg four times daily
  29-60 kg (64-132 lbs): trimethoprim-sulfamethoxazole 80/400 mg four times daily
  60 kg (132 lbs): trimethoprim-sulfamethoxazole 80/400 mg four times daily
  60-80 kg (132-176 lbs): trimethoprim-sulfamethoxazole 160/800 mg three times daily
  > 80 kg (176 lbs): trimethoprim-sulfamethoxazole 160/800 mg four times daily
  Other Names: Bactrim; Co-trimoxazole; Septra
  Arms: Standard plus anti-CA-MRSA
Drug: Cephalexin — Weight-based dosing in capsule or suspension form according to the following scale:
  15-19 kg (33-42 lbs): Cephalexin 300 mg four times daily
  20-24 kg (42-53 lbs): Cephalexin 400 mg four times daily
  25-29 kg (53-64 lbs): Cephalexin 500 mg four times daily
  29-60 kg (64-132 lbs): Cephalexin 500 mg four times daily
  60-80 kg (132-176 lbs): Cephalexin 1000 mg three times daily
  > 80 kg (176 lbs): Cephalexin 1000 mg four times daily
  Other Names: Keflex

SUMMARY:
The primary aim of this study is to quantify the effectiveness of Bactrim as additional therapy for the treatment of uncomplicated cellulitis in adults, by comparing: standard therapy plus Bactrim, versus standard therapy plus placebo.

The primary hypothesis of this study is that, in light of increasing CA-MRSA prevalence, subjects treated with standard therapy plus Bactrim will have higher cure rates than those treated with standard therapy plus placebo.

ELIGIBILITY:
Inclusion Criteria

* Must have cellulitis as defined here:

  1. Definition A (preferred definition):

     Recent onset of soft tissue erythema, considered by the treating clinician to be bacterial in origin, and associated with signs of infection that include at least two of the following: pain, swelling, warmth, fever, lymphangitis, induration, or ulceration.
  2. Definition B (ONLY for darkly-pigmented subjects who cannot use Definition A):

     Recent onset of soft tissue color change, pain, or swelling, considered by the treating clinician to be bacterial in origin, and at least one of the following: warmth, fever, induration, or ulceration
* Clinical (non-research) attending physician agrees with treatment with cephalexin until 3 days after all symptoms gone, using our weight-based dosing
* Responsible clinical attending physician comfortable with adding trimethoprim-sulfamethoxazole vs. placebo to the above
* Subject understands the study and signs written informed consent.
* Subject agrees to drink at least 1 liter of fluid per day.
* Subject will commit to all follow-up appointments

Exclusion Criteria:

* Age < 12 months or weight <15 kg
* Current skin infection has already been treated
* Allergy to sulfa drugs
* History of severe allergic reaction to penicillin (defined as anaphylactoid reaction, angioedema, bronchospasm)
* Current use of any antibiotic (other than topicals)
* Diabetes mellitus
* Cellulitis complicated by underlying peripheral vascular disease
* Renal insufficiency, defined as patient report, clinical suspicion, or creatinine>1.3 or EGFR<60 on the last-available set of chemistry results in our computer system
* Hospital admission required
* Presence of > 1 cc of purulent discharge at any time
* Cellulitis involving an indwelling vascular, enteric, or urinary catheter
* Immunocompromise of any etiology
* Pregnancy
* Breast feeding
* Facial cellulitis (infection is above the clavicles)
* Cellulitis associated with marine or freshwater injury, or animal or human bite. (Insect bites not excluded.)
* History of glucose-6-phosphate dehydrogenase deficiency
* Taking coumadin (warfarin), methotrexate, cisapride, phenytoin (dilantin), digoxin, or dofetilide
* Known megaloblastic anemia due to folate deficiency.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2007-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Pallin, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts

REFERENCES:
- [Derived] Pallin DJ, Binder WD, Allen MB, Lederman M, Parmar S, Filbin MR, Hooper DC, Camargo CA Jr. Clinical trial: comparative effectiveness of cephalexin plus trimethoprim-sulfamethoxazole versus cephalexin alone for treatment of uncomplicated cellulitis: a randomized controlled trial. Clin Infect Dis. 2013 Jun;56(12):1754-62. doi: 10.1093/cid/cit122. Epub 2013 Mar 1. PMID 23457080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled generally-healthy subjects with uncomplicated acute cellulitis from 6/2007 to 12/2011. Eligible subjects were adults and children presenting to EDs of 3 teaching hospitals in Boston, MA.
Pre-assignment Details: Each subject was assigned randomly to a treatment group by the institutions' research pharmacies. The research pharmacies had no knowledge of subjects' clinical characteristics. Treating (non-research) clinicians, research clinicians, coordinators, and subjects had no knowledge of the randomization sequence.
Groups:
- Trimethoprim-sulfamethoxazole: Cephalexin plus trimethoprim-sulfamethoxazole
- Placebo: Cephalexin plus placebo
Period: Overall Study
Arm/Group | Trimethoprim-sulfamethoxazole | Placebo
Started | 76 | 77
Completed | 73 | 73
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Found ineligible | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trimethoprim-sulfamethoxazole | Placebo | Total
Number analyzed (Participants) | 76 | 77 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 5 | 8
  Between 18 and 65 years | 68 | 69 | 137
  >=65 years | 5 | 3 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 37.03 (15.07) | 32.43 (15.15) | 34.71 (15.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 36 | 75
  Male | 37 | 41 | 78
Region of Enrollment [Number; unit: participants]
  United States | 76 | 77 | 153

OUTCOME MEASURES:

1. Primary Outcome: Relative Efficacy
Description: Proportion of subjects in each arm with successful treatment.
  Treatment success was assessed by physician examination at 12 +/- 2 days. Non-success was defined as subsequent hospitalization, change in antibiotics, surgical or needle drainage of an abscess, or recurrence of infection within 30 days. Cure was defined as resolution of all symptoms other than mild residual erythema or edema. We confirmed the determination of cure by telephone interview and medical record review at 30 +/- 2 days.
Time Frame: 12 +/- 2 days; 30 +/- 2 days
Population: Of the 153 randomized subjects, 4 were randomized in error and did not receive study drug, 1 received two doses before it was discovered that he was ineligible, 1 was lost to follow up, and 1 withdrew voluntarily in the first few days after enrollment. This left 146 subjects for intent-to-treat analysis.
Measure: Number; unit: participants
Arm/Group | Trimethoprim-sulfamethoxazole | Placebo
Number analyzed (Participants) | 73 | 73
participants | 62 | 60
Statistical Analysis 1: Comparison: Trimethoprim-sulfamethoxazole vs Placebo; The study was powered to detect a difference in cure rate of 98% in the intervention group vs. 85% in the control group, with 2-sided alpha 0.05. This would yield a number needed to treat of 7.7 for intervention vs. control, and required 144 subjects to achieve 80% power. No data were analyzed until study completion; Test type: Superiority or Other; p < 0.05, Chi-squared; Risk Difference (RD) = 2.7, 95% CI [-9.3 to 15]

2. Secondary Outcome: Progression to Abscess
Description: Proportion of subjects in each arm with progression from cellulitis to abscess.
Time Frame: 12 +/- 2 days, 30 days +/- 2 days
Measure: Number; unit: participants
Arm/Group | Trimethoprim-sulfamethoxazole | Placebo
Number analyzed (Participants) | 73 | 73
participants | 5 | 5
Statistical Analysis 1: Comparison: Trimethoprim-sulfamethoxazole vs Placebo; We assessed the rate of progression to abscess in the two groups; Test type: Superiority or Other; p < 0.05, Chi-squared; Risk Difference (RD) = 0, 95% CI 2-sided [-6.5 to 6.3]

ADVERSE EVENTS:
Time Frame: 30 days, assessed via telephone contact, in-person visit, and medical record review.
Description: Serious adverse events were considered to be those resulting in hospital admission.
Arm/Group | Trimethoprim-sulfamethoxazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/73 | 1/73
Other Adverse Events (participants affected / at risk) | 36/73 | 39/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trimethoprim-sulfamethoxazole (N=73) | Placebo (N=73)
Clostridium difficile colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trimethoprim-sulfamethoxazole (N=73) | Placebo (N=73)
Diarrhea (Gastrointestinal disorders) | 21 | 25
Vomiting (Gastrointestinal disorders) | 5 | 8
Nausea (Gastrointestinal disorders) | 15 | 13
Pruritis (Skin and subcutaneous tissue disorders) | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes